CLINICAL TRIAL: NCT06002217
Title: Echo-guided Transverse Abdominal Plane Block (TAP) in Anterior Lumbar Arthrodesis (ALIF): Randomized, Double-blind, Controlled Trial.
Brief Title: Echo-guided Transverse Abdominal Plane Block (TAP) in Anterior Lumbar Arthrodesis (ALIF)
Acronym: TAP ALIF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Guillaume LONJON, Principal investigator, Clinique Saint Jean, France
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A00970-43
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Fusion of Spine, Lumbar Region
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Active Comparator)
  Interventions: Drug: Levobupivacaine
- saline solution (Placebo Comparator)
  Interventions: Other: Placebo Tap block

INTERVENTIONS:
Drug: Levobupivacaine — Patients in the tap block arm will receive an injection of levobupivacaine 2.5mg/ml
  Arms: TAP Block
Other: Placebo Tap block — Patients in the placebo arm will receive an injection of salin solution 2.5mg/ml , in the same way as tap block
  Arms: saline solution

SUMMARY:
The goal of this interventional study is to is to compare the effect of a tap block versus a placebo in patients undergoing anterior lumbar spine surgery.

The main question it aims to answer :

• whether tap block can reduce the need for postoperative pain medication Participants will be randomized into two groups and all postoperative pain medication will be recorded over 3 days.

Researchers will compare tap block vs placebo to see if it reduces postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

Patient affiliated or entitled to a social security plan.

* Patient who has been informed about the study and has co-signed a consent form with the investigator. consent to participate in the study.
* Patients over 18 years of age scheduled for abdominal disc surgery on one or two levels.
* Patient with ASA criteria 1, 2 and 3.

Exclusion Criteria:

* Patients with intolerance or contraindication to paracetamol, anti-inflammatory or morphine.
* Patients allergic to local anesthetics.
* Pregnant or breast-feeding patient.
* patient undergoing cancer or trauma surgery trauma.
* Patient participating in another interventional study.
* Patient with a history of lumbar arthrodesis.
* Patient refusing to sign consent form.
* Patient unable to give informed consent.
* Patient under court protection, guardianship or trusteeship.
* Patient not available for study follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | 72hours
  The use of analgesics (oral or venous) during the during the 72 hours following surgery

SECONDARY OUTCOMES:
Pain assessment will be reported for 72 hours after surgery measured on a Visual analogue scale between 0 and 10 | 72hours
  Pain assessment for 72 hours after surgery, measured on a scale between 0 and 10 (VAS scale ), where 0 is no pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St jean sud de france, Montpellier, France

IPD SHARING:
Plan to Share IPD: No